CLINICAL TRIAL: NCT05782595
Title: BODY BALANCE RESPONSES TO AQUATIC THERAPY AMONG ACOHORT OF HEALTHY POSTMENOPAUSAL WOMEN
Brief Title: Body Balance Responses to Aquatic Therapy Among a Cohort of Healthy Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Mabrouk Ali, BODY BALANCE RESPONSES TO AQUATIC THERAPY AMONG ACOHORT OF HEALTH POSTMENOPAUSAL WOMEN, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012/003731
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Postmenopausal Women
Keywords: Aquatic therapy
MeSH Terms: interventions — Aquatic Therapy; Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Aquatic therapy
Masking Description: Randome generator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquatic therapy (Experimental): Aquatic exercise program: Each woman in group (A) will receive aquatic exercises for 40 minutes.
  Interventions: Other: Aquatic therapy

INTERVENTIONS:
Other: Aquatic therapy — • Each session was divided into three phases:
  1. Aquatic environment adaptation phase
  2. stretching phase
  3. a phase of static and dynamic exercises for balance
  Other Names: Hydrotherapy

SUMMARY:
the aim of this study is to investigate the effect of aquatic Exercises on balance in healthy postmenopausal women .

DETAILED DESCRIPTION:
Menopause, defined as the final menstrual period, physiologically results from the natural depletion of ovarian follicular function; a condition that translates into permanent amenorrhea (the permanent cessation of menstrual flow) generally associated with aging.

Many women have few or no symptoms, and thus, these women are not necessarily in need of medical treatment. The signs and symptoms of menopause are characterized by onset of irregular menses, hot flushes and night sweats. Menopause is also known to be associated with changes in behavior and other biological functions e.g., mood swings, anxiety, stress, forgetfulness and sleep disturbances

ELIGIBILITY:
Inclusion Criteria:

* 1) Their ages will range from 50 to 60 years.

  2) Their BMI will be less than 30 kg/m².

  3) All females will be apparently healthy postmenopausal women and walking independency.

  4) They have physical ability to participate in aquatic exercise program.

Exclusion Criteria:

* 1)Urinary or fecal incontinence. 2)Open wounds, contagious skin diseases or infective diseases. 3) Vascular thrombi. 4) Cardiac insufficiency. 5) Fracture in last year in lower limb.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Biodex balance assessment | 3 months
  It is objective device that measure dynamic postural stability and it is reliable for evaluating dynamic postural balance in healthy subjects

SECONDARY OUTCOMES:
The Timed Up and Down Stair Test | 3 months
  • This test is designed to measure dynamic balance (Leroux, 2005). Using an 8-inches high stair, the women will be asked to step on and off seven times at their naturally preferred comfortable pace. They step up with one foot and then the other and step down with one foot followed by the other foot.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mabrouk, Principal Investigator — faculty of physical therapy
Locations (1):
- Hala mabrouk ali, Giza, Egypt